CLINICAL TRIAL: NCT04660357
Title: Do Activity-Specific Balance Confidence and Fear of Fall Affect Autonomy and Social Participation in Individuals With Knee Osteoarthritis Above 65 Years Old?
Brief Title: Osteoarthritis, Balance, and Fear of Falling
Acronym: OA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Özgü İnal, principal investigator, Hacettepe University
Other Study IDs: 2020/281
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis | interventions — Longitudinal Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: survey study — survey study

SUMMARY:
Osteoarthritis (OA) is a progressive and irreversible degenerative joint disease characterized by marginal bone hypertrophy, erosion, and subchondral sclerosis in the articular cartilage.It has been determined that being of advanced age and joint involvement due to osteoarthritis are a risk factor for addiction in activities and this increases the individual's self-care ability and dependency in daily living activities.Older individuals with knee osteoarthritis may be at risk of falling.This study was planned to examine the relationship between activity-specific balance confidence and fear of falling, autonomy and social participation in individuals with knee osteoarthritis over 65 years of age.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a progressive and irreversible degenerative joint disease characterized by marginal bone hypertrophy, erosion, and subchondral sclerosis in the articular cartilage.It has been determined that being of advanced age and joint involvement due to osteoarthritis are a risk factor for addiction in activities and this increases the individual's self-care ability and dependency in daily living activities.Older individuals with knee osteoarthritis may be at risk of falling.Considering the relationship between the concepts of osteoarthritis and old age with the common concepts of daily life activity problems, falling, loss of autonomy and affecting social participation; this study was planned to examine the relationship between activity-specific balance confidence and fear of falling, autonomy and social participation in individuals with knee osteoarthritis over 65 years of age.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old
* Diagnosed with knee osteoarthritis according to ACR diagnostic criteria

Exclusion Criteria:

Not having enough cooperation

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: * 65 years old
  * Diagnosed with knee osteoarthritis according to ACR diagnostic criteria
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2021-09-20 (Estimated)

PRIMARY OUTCOMES:
WOMAC, The Activities-specific Balance Confidence Scale, Falls Efficacy Scale, The functional autonomy measurement system, Community Integration Questionnaire, Berg Balance Scale | 1 year
  The WOMAC index is a disease-specific, self-administered questionnaire developed to study patients with hip or knee OA. It consists of 24 questions, grouped into 3 subscales.Higher scores indicate more or worse symptoms, maximal limitations, and poor health.

CONTACTS AND LOCATIONS:
Overall Officials: Özgü İnal, Principal Investigator — Trakya University
Locations (1):
- Özgü İnal, Edirne, Merkez, Turkey (Türkiye)